CLINICAL TRIAL: NCT04079166
Title: A Phase 2, Multicentre, Open-Label, Umbrella Study of SCIB1 and iSCIB1+ in Patients With Advanced Unresectable Melanoma Receiving Nivolumab With Ipilimumab or SCIB1 With Pembrolizumab (The SCOPE Study)
Brief Title: SCIB1 and iSCIB1+ in Melanoma Patients Receiving Nivolumab With Ipilimumab or SCIB1 With Pembrolizumab (The SCOPE Study)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scancell Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCIB1-002
Record Dates: First submitted 2019-08-16; First posted 2019-09-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma; Melanoma (Skin); Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Open label, uncontrolled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCIB1 or iSCIB1+ (Experimental): SCIB1 or iSCIB1+ administered by needle-free injection
  Interventions: Biological: SCIB1 or iSCIB1+ DNA vaccine

INTERVENTIONS:
Biological: SCIB1 or iSCIB1+ DNA vaccine — Participants receive up to 11 doses of either SCIB1 or iSCIB1+ up to 85 weeks, in combination with nivolumab with ipilimumab or SCIB1 with pembrolizumab.
  Nivolumab with ipilimumab or pembrolizumab treatment will be started 1 week after the first dose of SCIB1 or iSCIB1+ and given as per standard treatment.

SUMMARY:
The purpose of this study is to find out if two new treatment cancer vaccines called SCIB1 and iSCIB1+ can be used safely when added to nivolumab (Opdivo) with ipilimumab (Yervoy), or SCIB1 with pembrolizumab (Keytruda). Pembrolizumab or nivolumab with ipilimumab are standard treatments approved for patients with advanced melanoma (skin cancer).

The study will also look to see if SCIB1 or iSCIB1+ can increase the likelihood that melanoma patients will respond to the standard treatments, and also if SCIB1 and iSCIB1+ can help to make those responses last longer. SCIB1 and iSCIB1+ are considered experimental. SCIB1 has been given to melanoma patients in an earlier study. It was generally well-tolerated, and researchers saw some signs that it may help to stimulate the immune system, which is a way in which the body can fight the cancer. iSCIB1+ is similar to SCIB1 but might benefit more patients with melanoma.

DETAILED DESCRIPTION:
This is an open label, single arm Phase 2 study to determine the response rate and safety and tolerability of SCIB1 or iSCIB1+ when added to nivolumab (Opdivo) with ipilimumab (Yervoy) or SCIB1 with pembrolizumab (Keytruda). Pembrolizumab or nivolumab with ipilimumab are standard treatments already approved for the treatment of advanced melanoma.

The plan for this study is for SCIB1 or iSCIB1+ to be given up to 11 times for 85 weeks, in combination with nivolumab with ipilimumab or SCIB1 with pembrolizumab. The standard treatments will be given according to the current label. The SCIB1 or iSCIB1+ injection will be given using PharmaJet needle-free injection device systems in the upper arm or upper leg.

Before treatment starts and after consent has been given, all patients will undergo screening tests (to be completed within 28 days of treatment initiation) to ensure the patient is eligible to take part. Over the 85-week treatment period, the patient will visit the hospital multiple times and have some telephone/video calls. The evaluations and procedures that will be carried out at each visit are all detailed in the study information sheets given to the patient before consent is taken.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of unresectable Stage III or Stage IV melanoma.
2. Not received prior systemic treatment for advanced disease. Prior neoadjuvant or adjuvant treatment, defined as treatment prior to or following resection of all detectable disease, is permitted; last dose must be at least 24 weeks before the first dose of SCIB1 or iSCIB1+.
3. Checkpoint inhibition with either nivolumab with ipilimumab or pembrolizumab will be an appropriate treatment for their advanced disease.
4. BRAF status must be known; patients with BRAF mutation positive disease may be enrolled without BRAF inhibitor treatment at the discretion of the Investigator, provided that they have no evidence of rapidly progressing disease.
5. At least one measurable lesion per RECIST 1.1 criteria by CT scan or MRI.
6. Human leukocyte antigen (HLA)-A2 positive (applicable for cohort 1, 2 and 3).
7. Positive for HLA-DR4, HLA-DR7, HLA-DR53 or HLA-DQ6 (applicable for cohort 1, 2 and 3).
8. Patients for whom nivolumab with ipilimumab is determined to be an appropriate treatment will be treated in cohort 4 with iSCIB1+ if:

   1. the target HLA haplotype does not match as stated in criteria number 6 and 7, or
   2. they are unable to wait for HLA screening results prior to enrolment or starting treatment, or
   3. cohort 1 and cohort 3 have completed or closed to recruitment.
9. At least 18 years of age.
10. A life expectancy of more than 3 months.
11. ECOG performance status of 0 or 1.
12. Adequate organ function as determined by protocol laboratory values.
13. Able and willing to provide written informed consent prior to any study related procedure.
14. Women of child-bearing potential must have a negative serum pregnancy test during screening and be neither breastfeeding nor intending to become pregnant during study participation, and shall be warned of potential foetal harm from nivolumab with ipilimumab or pembrolizumab. Women of child-bearing potential must agree to use highly effective contraceptive methods prior to study entry, for the whole duration of study treatment, and for 120 days after discontinuation of SCIB1 or iSCIB1+, or nivolumab with ipilimumab, or pembrolizumab, whichever is last.
15. Men who are potentially fertile with partners of childbearing potential must agree to use highly effective contraceptive methods for the whole duration of study treatment, and for 120 days after discontinuation of SCIB1 or iSCIB1+, or nivolumab with ipilimumab, or pembrolizumab, whichever is last.
16. Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. A diagnosis of mucosal, acral or ocular melanoma.
2. Has central nervous system metastases or carcinomatous meningitis.
3. Has previously received a treatment to block cytotoxic T lymphocyte associated protein 4 (CTLA-4), programmed cell death protein 1 (PD-1), PD-L1, or programmed death-ligand 2 (PD-L2) with the following exception: patients who have received neoadjuvant or adjuvant treatment with these treatments are eligible, provided that the last dose was administered at least 24 weeks before the first dose of SCIB1 or iSCIB1+.
4. Patients with lactate dehydrogenase (LDH) > 2 x ULN.
5. Expected to require any other form of systemic or localized anticancer therapy while receiving study treatment.
6. Taking any systemic steroid therapy within 1 week of the first dose of study drug or is receiving any other form of immune suppressant medication. Physiological doses of systemic steroids such as those for the management of adrenal insufficiency, as well as topical and inhaled steroids, such as those for the management of asthma, are permitted.
7. Receiving treatment with any investigational product within 28 days (or 5 half-lives of the treatment concerned) prior to the first dose of study treatment.
8. Has a previous (within 5 years) or current malignancy with the exception of melanoma, and curatively treated local tumours.
9. Has a concurrent illness which would preclude study conduct and assessment.
10. Has New York Heart Association class III or IV heart disease, myocardial infarction within previous 6 months, a heart rate of ≤ 50 beats per minute, a history of significant cardiac abnormality and/or clinically significant abnormal baseline ECG reading, active ischemia, or any other uncontrolled cardiac condition.
11. Has a history of severe hypersensitivity reaction to treatment with a monoclonal antibody.
12. Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents (patients with vitiligo or resolved childhood asthma/atopy are an exception and are not excluded for these conditions). The following patients are not excluded from the study: patients who require intermittent use of bronchodilators or local steroid injections, patients with hypothyroidism stable on hormone replacement, and patients who receive physiological doses of steroids as replacement therapy, such as those for the management of adrenal insufficiency. In such cases the recruiting investigator should discuss the patients' eligibility with the study Medical Monitor prior to enrolment.
13. Received a live vaccine within the 28 days prior to first dose of study treatment, or patient has received a non-live vaccine, including COVID-19 vaccines, within 14 days prior to first dose of study treatment.
14. A known history of human immunodeficiency virus (HIV) or has any positive test for hepatitis B virus or hepatitis C virus indicating active acute or chronic infection.
15. A known current or recent history (within the last year) of substance abuse including illicit drugs or alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessed by the evaluation of adverse events (AEs) (Run-In Sub-Cohorts) | Up to 30 days after the final dose of study drug
  National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events; CTCAE v5.0.
Safety and tolerability assessed by the evaluation of vital signs, physical examination, 12-lead ECG, laboratory assessments, performance status, injection site reaction and the use of concomitant medications (Run-In Sub-Cohorts) | Up to 30 days after the final dose of study drug
Objective response rate (ORR) (Main Study) | Up to 2 years (Week 97) from the first dose of study drug
  ORR assessed by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) criteria.

SECONDARY OUTCOMES:
Duration of response (Main Study) | Up to 2 years (Week 97) from the first dose of study drug
  Duration of response, measured from the point of first response (complete response or partial response) to the date of disease progression (per RECIST 1.1) or death due to any cause.
ORR assessed by the modified RECIST 1.1 for immune-based therapeutics (iRECIST) (Main Study) | Up to 2 years (Week 97) from the first dose of study drug
  ORR assessed by iRECIST criteria.
Progression Free Survival (PFS) rate | Up to 2 years (Week 97) from the first dose of study drug
  PFS rate is defined as the proportion of participants who have not progressed (per RECIST 1.1 and iRECIST), or started new anticancer therapy, or died.
Overall survival (OS) rate | Up to 2 years (Week 97) from the first dose of study drug
  OS rate is defined as the proportion of participants who remain alive.
Safety and tolerability by the evaluation of AEs (Main Study) | Up to 30 days after the final dose of study drug
  NCI CTCAE v5.0.
Safety and tolerability by the evaluation of vital signs, physical examination, 12-lead ECG, laboratory assessments, performance status, injection site reaction and the use of concomitant medications (Main Study) | Up to 30 days after the final dose of study drug

OTHER OUTCOMES:
Exploratory: Immune response | Up to 30 days after the final dose of study treatment
  Immune response as measured using ELISpot and other assays on peripheral blood samples from patients.
Exploratory: Marker expression | Up to 30 days after the final dose of study treatment
  Analysis of tumour biopsy samples for various markers.

CONTACTS AND LOCATIONS:
Overall Officials: Poulam Patel, Principal Investigator — University of Nottingham
Locations (15):
- United Kingdom (15):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre University NHS Trust, Cardiff
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - East and North Hertfordshire NHS Trust, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospital NHS Foundation Trust, Oxford
  - University Hospital Plymouth NHS Trust, Plymouth
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.